CLINICAL TRIAL: NCT02310477
Title: REBECCA: A Cohort Study of Regorafenib in the Real-life Setting in Patients Previously Treated for Metastatic Colorectal Cancer.
Brief Title: Regorafenib in Metastatic Colorectal Cancer : a Cohort Study in the Real-life Setting
Acronym: REBECCA
Status: Completed | Type: Observational
Sponsor: Centre Oscar Lambret (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: REBECCA-1305
Record Dates: First submitted 2014-10-08; First posted 2014-12-08 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-01

CONDITIONS: Metastatic Colorectal Cancer
Keywords: regorafenib, cohort, metastatic colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — regorafenib

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: regorafenib — regorafenib for all groups
  Other Names: stivarga

SUMMARY:
This is a largest cohort study aimed to estimate the overall survival of patients been treated with regorafenib for metastatic colorectal cancer (mCRC) within the frame of a french compassionate program.

DETAILED DESCRIPTION:
Regorafenib (REG) is a multi-kinase inhibitor with survival benefits in patients with pretreated mCRC, as demonstrated in the phase III CORRECT study. As a result, REG has been made available for medical practice use in the US, and in the Europe. However, prescribing conditions in the real-life setting are known to be less stringent than selection criteria in clinical trials. The REgorafeniB in mEtastatic Colorectal cancer: a French Compassionate progrAm (REBECCA) is an ambispective cohort study designed to elucidate safety and effectiveness outcomes associated with REG as used in clinical practice for mCRC who have been previously treated with, or are not considered candidates for, available therapies.

Patients were identified from the database of the French ATU (Temporary Authorization for Use), approved by the French Health Authorities to provide early access to innovative, not yet approved medicinal products such as REG.

Baseline patient and tumor characteristics, REG dosing and dose-intensity, REG-related adverse events, pre- and post REG treatments, predictors of events, and effectiveness data (PFS, OS) were collected from patients who agreed, and whom physicians accepted to collaborate on the REBECCA cohort.

ELIGIBILITY:
Inclusion criteria :

* Patient ≥ 18 years old
* With a colorectal cancer metastatic histologically proven
* Have met the criteria defined in the monograph ATU (Temporary Authorization for Use) validated by French Health Authorities and for which the request for access to treatment has been validated, that is in patients with mCRC as used in clinical practice for mCRC who have been previously treated with, or are not considered candidates for, available therapies.
* Patients who received at least one dose on REG

Exclusion criteria :

* Opposed to the study
* Patient does not meet the inclusion criteria
* Patient deprived of liberty or under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were identified from the database of the French ATU (Temporary Authorization for Use), approved by the French Health Authorities to provide early access to innovative, not yet approved medicinal products such as REG.
  elligible patients were those who accepted to participate to the cohort study, and whom physicians accepted to collaborate on the REBECCA cohort.
Sampling Method: Non-Probability Sample
Enrollment: 704 (Actual)
Dates: Start 2014-02; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | at death or at the end of study
  median time between the date of the first administration REG and the date of the death

SECONDARY OUTCOMES:
Patients and tumor baseline characteristics | at the end of treatment
  Tumor location, KRAS status, synchronous or metachronus metastases, time elapsed from diagnosis of metastases, surgery of the primary, previous times of treatment, weight/height/BMI, ECOG, met location, age, performance status
Time under REG treatment | at the end of treatment
  calculated from the start of treatment until the treatment discontinuation for any cause) and within some subgroups of patients:Tumor location, KRAS status, synchronous or metachronus metastases, time elapsed from diagnosis of metastases, surgery of the primary, previous times of treatment, weight/height/BMI, ECOG, met location, age, performance status, initial REG dosage
Compliance | at the end of study
  dose-intensity of treatment with REG, including the actual daily dosage
Safety of REG | at the end of treatment
  according to NCI-CTCAE (Common Toxicity Criteria for Adverse Effects) v4.0 and within some subgroups of patients
Potential predictive factors | at the end of study
  regarding tolerance, time under REG treatment, PFS, and OS.
Progression-free survival (PFS) | at the end of study
  median time between the date of the first administration REG and the date of the first progression

CONTACTS AND LOCATIONS:
Overall Officials: Antoine ADENIS, MD, Principal Investigator — Centre Oscar Lambret
Locations (1):
- Centre Oscar Lambret, Lille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adenis A, de la Fouchardiere C, Paule B, Burtin P, Tougeron D, Wallet J, Dourthe LM, Etienne PL, Mineur L, Clisant S, Phelip JM, Kramar A, Andre T. Survival, safety, and prognostic factors for outcome with Regorafenib in patients with metastatic colorectal cancer refractory to standard therapies: results from a multicenter study (REBECCA) nested within a compassionate use program. BMC Cancer. 2016 Jul 7;16:412. doi: 10.1186/s12885-016-2440-9. PMID 27389564